CLINICAL TRIAL: NCT06317974
Title: The Effect of Breastfeeding Education Based on the Health Belief Model Given ın the Third Trimester of Pregnancy on Couples Breast Milk Perception and Self-efficacy
Brief Title: The Effect of Breastfeeding Education on Breast Milk Perception and Self-Efficacy in the Pregnancy Health Belief Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Leman Yılmaz Cesur, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/210
Record Dates: First submitted 2024-01-04; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Breastfeeding Education
Keywords: Health Belief Model; Breastfeeding Self-Efficacy; Breast milk; Breastfeeding; Parent education
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized controlled, experimental research design in pre-test, post-test design Made with
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Breastfeeding education was given to the intervention group based on the health belief model.
  Interventions: Behavioral: Breastfeeding education based on the Health Belief model
- control group (No Intervention): The control group received standard care.

INTERVENTIONS:
Behavioral: Breastfeeding education based on the Health Belief model — Training was given face to face with the participant, lasting approximately 40 minutes. One week after the training presentation, three short messages about the training were sent to the couples (both the pregnant woman and her partner) every other day. Two weeks after the training was given, a phone call was made for feedback. Post-test data were taken four weeks later.
  Arms: Intervention group

SUMMARY:
Objective: The aim of this study was to evaluate the effect of breastfeeding education based on the Health Belief Model during the antenatal period on couples' perception and self-efficacy regarding breast milk.

DETAILED DESCRIPTION:
Introduction: It is known that breast milk is crucial for newborns and infants. The Health Belief Model has been widely used in recent years to improve and promote health behaviors.

Objective: The aim of this study was to evaluate the effect of breastfeeding education based on the Health Belief Model during the antenatal period on couples' perception and self-efficacy regarding breast milk.

Method: This randomized controlled study was conducted between June 30, 2022, and December 31, 2022, at the Dr. Selahattin Cizrelioğlu State Hospital in Şırnak. A total of 220 participants, including 110 couples who met the inclusion criteria, were randomly assigned to an intervention group (55 couples) and a control group (55 couples). Data were collected using a "Participant Information Form" for socio-demographic and obstetric information, the "Adults' Perception of Breast Milk Scale" for assessing perception related to breast milk, the "Pregnancy Breastfeeding Self-Efficacy Scale- Short Form" for evaluating mothers' breastfeeding self-efficacy during the antenatal period, and the "Paternal Breastfeeding Self-Efficacy Scale" for assessing fathers' breastfeeding self-efficacy during the pregnancy period.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18 and over
* Living in the same house with his/her spouse
* Able to speak and understand Turkish
* In the 27th week of pregnancy and above
* Having a first pregnancy
* Using a phone
* Couples willing to participate in the research

Exclusion Criteria:

* multiparous
* Receiving psychiatric or neurological treatment that affects cooperation and cognitive functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Mothers' and fathers' perception of breast milk, assessed using the Adults' Breast Milk Perception Scale. | 30 days
  In this study, it was determined that breastfeeding education given based on the health belief model in the last trimester of pregnancy increased the breast milk perception levels of expectant mothers and fathers.

SECONDARY OUTCOMES:
Breastfeeding self-efficacy of mothers evaluated using the Breastfeeding Self-Efficacy Scale-Short Form during Pregnancy | 30 days
  In this study, it was determined that breastfeeding education given in the pregnancy health belief model increased pregnant women's breastfeeding self-efficacy levels during pregnancy.

OTHER OUTCOMES:
Paternal breastfeeding self-efficacy assessed using the Paternal Breastfeeding Self-Efficacy Scale. | 30 days
  In this study, it was determined that breastfeeding education given in the health belief model during pregnancy increased fathers' breastfeeding self-efficacy levels.

CONTACTS AND LOCATIONS:
Overall Officials: Leman Yılmaz Cesur, Principal Investigator — Msc Midwife
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dror DK, Allen LH. Overview of Nutrients in Human Milk. Adv Nutr. 2018 May 1;9(suppl_1):278S-294S. doi: 10.1093/advances/nmy022. PMID 29846526
- [Background] Alex A, Bhandary E, McGuire KP. Anatomy and Physiology of the Breast during Pregnancy and Lactation. Adv Exp Med Biol. 2020;1252:3-7. doi: 10.1007/978-3-030-41596-9_1. PMID 32816256
- [Background] Ballard O, Morrow AL. Human milk composition: nutrients and bioactive factors. Pediatr Clin North Am. 2013 Feb;60(1):49-74. doi: 10.1016/j.pcl.2012.10.002. PMID 23178060
- [Background] Boix-Amoros A, Collado MC, Van't Land B, Calvert A, Le Doare K, Garssen J, Hanna H, Khaleva E, Peroni DG, Geddes DT, Kozyrskyj AL, Warner JO, Munblit D. Reviewing the evidence on breast milk composition and immunological outcomes. Nutr Rev. 2019 Aug 1;77(8):541-556. doi: 10.1093/nutrit/nuz019. PMID 31111150
- [Background] Ceriani Cernadas JM. Colostrum and breast milk in the neonatal period: The benefits keep adding up. Arch Argent Pediatr. 2018 Aug 1;116(4):234-235. doi: 10.5546/aap.2018.eng.234. No abstract available. English, Spanish. PMID 30016015
- [Background] Chen S, Li L, Sun Q, Chen S, Cheng J, Xiong S. Effect of IMB Model Combined with Spousal Support Breastfeeding Intervention on PBSES Score and Breastfeeding Rate of Primipara with Chronic Hepatitis B Virus Infection. Biomed Res Int. 2022 Sep 15;2022:9661408. doi: 10.1155/2022/9661408. eCollection 2022. PMID 36158886
- [Background] Dagla C, Antoniou E, Sarantaki A, Iliadou M, Mrvoljak-Theodoropoulou I, Andersson E, Dagla M. The Effect of Antenatal Education on Expectant Fathers' Attitudes toward Breastfeeding and Attachment to the Fetus. Nurs Rep. 2023 Feb 12;13(1):243-254. doi: 10.3390/nursrep13010023. PMID 36810274
- [Background] Dennis CL, Faux S. Development and psychometric testing of the Breastfeeding Self-Efficacy Scale. Res Nurs Health. 1999 Oct;22(5):399-409. doi: 10.1002/(sici)1098-240x(199910)22:53.0.co;2-4. PMID 10520192
- [Background] Dennis CL, Brennenstuhl S, Abbass-Dick J. Measuring paternal breastfeeding self-efficacy: A psychometric evaluation of the Breastfeeding Self-Efficacy Scale-Short Form among fathers. Midwifery. 2018 Sep;64:17-22. doi: 10.1016/j.midw.2018.05.005. Epub 2018 May 15. PMID 29864577
- [Background] Correction to: ABM Clinical Protocol #8: Human Milk Storage Information for Home Use for Full-Term Infants, Revised 2017, by Eglash A, Simon L, and The Academy of Breastfeeding Medicine Breastfeed Med 2017;12(7):390-395. DOI: 10.1089/dna.2017.29047.aje. Breastfeed Med. 2018 Jul/Aug;13(6):459. doi: 10.1089/bfm.2017.29047.aje.correx. Epub 2018 Jun 29. No abstract available. PMID 29958002
- [Background] Hu L, Ding T, Hu J, Luo B. Promoting breastfeeding in Chinese women undergoing cesarean section based on the health belief model: A randomized controlled trial. Medicine (Baltimore). 2020 Jul 10;99(28):e20815. doi: 10.1097/MD.0000000000020815. PMID 32664074
- [Background] Kehinde J, O'Donnell C, Grealish A. The effectiveness of prenatal breastfeeding education on breastfeeding uptake postpartum: A systematic review. Midwifery. 2023 Mar;118:103579. doi: 10.1016/j.midw.2022.103579. Epub 2022 Dec 14. PMID 36580847
- [Background] Lumbiganon P, Martis R, Laopaiboon M, Festin MR, Ho JJ, Hakimi M. Antenatal breastfeeding education for increasing breastfeeding duration. Cochrane Database Syst Rev. 2016 Dec 6;12(12):CD006425. doi: 10.1002/14651858.CD006425.pub4. PMID 27922724
- [Background] Alus Tokat M, Okumus H, Dennis CL. Translation and psychometric assessment of the Breast-feeding Self-Efficacy Scale-Short Form among pregnant and postnatal women in Turkey. Midwifery. 2010 Feb;26(1):101-8. doi: 10.1016/j.midw.2008.04.002. Epub 2008 Jun 9. PMID 18541350
- [Result] Abuidhail J, Mrayan L, Jaradat D. Evaluating effects of prenatal web-based breastfeeding education for pregnant mothers in their third trimester of pregnancy: Prospective randomized control trial. Midwifery. 2019 Feb;69:143-149. doi: 10.1016/j.midw.2018.11.015. Epub 2018 Nov 28. PMID 30513445
- [Result] Atkinson L, Silverio SA, Bick D, Fallon V. Relationships between paternal attitudes, paternal involvement, and infant-feeding outcomes: Mixed-methods findings from a global on-line survey of English-speaking fathers. Matern Child Nutr. 2021 Jul;17 Suppl 1(Suppl 1):e13147. doi: 10.1111/mcn.13147. PMID 34241959
- [Result] Crippa BL, Consales A, Morniroli D, Lunetto F, Bettinelli ME, Sannino P, Rampini S, Zanotta L, Marchisio P, Plevani L, Gianni ML, Mosca F, Colombo L. From dyad to triad: a survey on fathers' knowledge and attitudes toward breastfeeding. Eur J Pediatr. 2021 Sep;180(9):2861-2869. doi: 10.1007/s00431-021-04034-x. Epub 2021 Mar 29. PMID 33779804
- [Result] Eaton L. Unwanted pregnancies fall worldwide but women in poorer countries remain disadvantaged, study finds. BMJ. 2020 Jul 24;370:m2985. doi: 10.1136/bmj.m2985. No abstract available. PMID 32709616
- [Result] Gebremariam KT, Zelenko O, Mulugeta A, Gallegos D. A cross-sectional comparison of breastfeeding knowledge, attitudes, and perceived partners' support among expectant couples in Mekelle, Ethiopia. Int Breastfeed J. 2021 Jan 4;16(1):3. doi: 10.1186/s13006-020-00355-z. PMID 33397410
- [Result] Han FL, Ho YJ, McGrath JM. The influence of breastfeeding attitudes on breastfeeding behavior of postpartum women and their spouses. Heliyon. 2023 Feb 23;9(3):e13987. doi: 10.1016/j.heliyon.2023.e13987. eCollection 2023 Mar. PMID 36879970
- [Result] Krikitrat P, Park CG, McCreary LL, Koenig MD, Abboud S, Sansiriphun N, Patil CL. Relationships between Thai fathers' self-efficacy to support breastfeeding and exclusive breastfeeding duration. Midwifery. 2022 Mar;106:103261. doi: 10.1016/j.midw.2022.103261. Epub 2022 Jan 19. PMID 35085913
- [Result] Liu L, Xiao G, Zhang T, Zhou M, Li X, Zhang Y, Owusua T, Chen Y, Qin C. Levels and Determinants of Antenatal Breastfeeding Attitudes among Pregnant Women: A Cross-Sectional Study. Children (Basel). 2023 Jan 31;10(2):275. doi: 10.3390/children10020275. PMID 36832403
- [Result] Naja F, Chatila A, Ayoub JJ, Abbas N, Mahmoud A; MINA collaborators; Abdulmalik MA, Nasreddine L. Prenatal breastfeeding knowledge, attitude and intention, and their associations with feeding practices during the first six months of life: a cohort study in Lebanon and Qatar. Int Breastfeed J. 2022 Feb 24;17(1):15. doi: 10.1186/s13006-022-00456-x. PMID 35209913
- [Result] Rabiepoor S, Khodaei A, Valizadeh R. Husbands' participation in prenatal care and breastfeeding self-efficacy in Iranian women: A randomized clinical trial. Med J Islam Repub Iran. 2019 Jun 20;33:58. doi: 10.34171/mjiri.33.58. eCollection 2019. PMID 31456982
- [Result] Titaley CR, Dibley MJ, Ariawan I, Mu'asyaroh A, Alam A, Damayanti R, Do TT, Ferguson E, Htet K, Li M, Sutrisna A, Fahmida U. Determinants of low breastfeeding self-efficacy amongst mothers of children aged less than six months: results from the BADUTA study in East Java, Indonesia. Int Breastfeed J. 2021 Jan 19;16(1):12. doi: 10.1186/s13006-021-00357-5. PMID 33468196
- [Result] Yakubu I, Garmaroudi G, Sadeghi R, Tol A, Yekaninejad MS, Yidana A. Assessing the impact of an educational intervention program on sexual abstinence based on the health belief model amongst adolescent girls in Northern Ghana, a cluster randomised control trial. Reprod Health. 2019 Aug 15;16(1):124. doi: 10.1186/s12978-019-0784-8. PMID 31416450
- [Result] Yavuz Donmez A, Korgali EU. The relationship between the perception of breast milk of parents with term infants and exclusive breastfeeding in the postnatal first six months. Turk Arch Pediatr. 2021 Jan 12;56(2):164-172. doi: 10.14744/TurkPediatriArs.2020.75875. eCollection 2021 Mar. PMID 34286328